CLINICAL TRIAL: NCT06598865
Title: Comparative Effectiveness on Glycemic Balance of a Non-pharmacological Treatment, Adapted Physical Activity (APA), Either Supervised by a Qualified APA Instructor or Unsupervised in Autonomy, in Individuals With Inadequately Controlled Type 2 Diabetes, Under Diet Alone or Non-insulin Treatment.
Brief Title: Comparative Effectiveness of Prescribed Adapted Physical Activity (APA), Either Practiced Independently After Training, or Supervised by an APA Teacher, on Glycemic Regulation in People With Unbalanced Type 2 Diabetes.
Acronym: ACTIDIAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A01320-47
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetes, Type 2; Non-Insulin Dependent; Poorly Controlled Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): after initial APA training, patients will be asked to implement APA sessions on their own for the duration of the study. They will then be asked to return to the investigating center for a visit at 3 months (Visit 3) to assess the effect of the APA carried out during this period.
- experimental (Experimental): after initial APA training, patients will receive regular support from an APA teacher, and will be asked to carry out 3 APA sessions a week, if possible in a Sport-Santé centre close to their home, for the duration of the study. The content of additional APA sessions (up to 2 additional sessions per week) can be discussed with the APA teacher.
  They will also be asked to return to the investigating center for a visit at 3 months (Visit 3) to assess the effect of the APA carried out during this period.
  Interventions: Other: adapted physical activity

INTERVENTIONS:
Other: adapted physical activity — After the initial training in adapted physical activity (APA), patients will receive regular support from an APA instructor, and they will be asked to participate in 3 sessions per week of APA, if possible in a Sport-Health center close to their home, for the entire duration of the study. The content of the additional APA sessions (up to 2 additional sessions per week) can be discussed with the APA instructor. They will also be asked to return to the study center for a visit at 3 months (Visit 3) to assess the effect of the APA conducted during this period
  Arms: experimental

SUMMARY:
Comparative effectiveness on glycemic balance of a non-pharmacological treatment, Adapted Physical Activity (APA), either supervised by a qualified APA instructor or unsupervised in autonomy, in individuals with inadequately controlled Type 2 Diabetes, under diet alone or non-insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given consent to participate in the study and has signed an informed consent form.
* Patient aged 18 to 67 years
* Patient diagnosed with type 2 diabetes
* Patient newly diagnosed or on non-insulin treatment (metformin +/- DPP4 inhibitor, GLP1 analogue +/- SGLT2 inhibitor) for whom it is considered to initiate or intensify antidiabetic treatment by introducing a new therapeutic class.
* Patient insufficiently controlled (> 1.30 g/L fasting blood glucose measured in the laboratory twice a few days apart in a city laboratory)
* Patient with good venous access.
* Patient capable of engaging in regular physical activity
* Patient who has undergone a coronary artery disease screening test in the year prior to inclusion according to the new recommendations of an expert consensus.
* Patient agrees to wear a FitBit Charge 6 bracelet for the entire duration of the study, including the run-in period, and agrees to recharge it and transmit the data.

Exclusion Criteria:

* Patient diagnosed with type 1 diabetes
* Patient treated with sulfonylureas
* Patient with a history of severe cardiovascular diseases (myocardial infarction, acute coronary syndrome, or stroke in the past year)
* Patient presenting a medical contraindication to performing a physical activity session (uncontrolled resting hypertension, i.e., systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg, unstable coronary artery disease, heart failure, severe proliferative or non-proliferative evolving retinopathy (unstabilized), or having undergone recent surgical laser treatment of the eye, plantar perforating ulcer, disabling osteoarthritis of the lower limbs, respiratory failure, severe renal impairment, liver failure, severe dysautonomia, i.e., risk of chronotropic insufficiency during exercise, peripheral neuropathy)
* Patient with a history of severe hypoglycemia in the 6 months prior to entering the study and/or not feeling their hypoglycemia at all
* Patient with an IPAQ score in the high category
* Patient with a known latex allergy
* Patient with morbid obesity (BMI > 40 kg/m²)
* Other conditions that may interfere with glycemic variation: particularly the use of corticosteroids during the study
* Patient treated with beta-blockers or calcium channel blockers with negative chronotropic action (such as isoptin)
* Breastfeeding woman
* Pregnant woman* or wishing to become pregnant

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of a 3-month re-training program, by comparing glycemic averages (measured for 10 consecutive days at 3 months, by a continuous glucose monitoring device (CGM) between experimental group (APA) vs control group. | 10 days after 3-month re-training program
  Measurement of glucose by CGM

CONTACTS AND LOCATIONS:
Locations (1):
- CERITD (Centre d'Etudes et de Recherches pour l'Intensification du Traitement du Diabète),, Évry, France

IPD SHARING:
Plan to Share IPD: No